CLINICAL TRIAL: NCT07047066
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of Flazoparib Combined With Temozolomide After the Completion of Standard Concurrent Chemoradiotherapy (CCRT) in Newly Diagnosed Glioblastoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Guangyuan Hu, Director, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBM-Ⅱ-001
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — fluzoparib; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib combined with Temozolomide (Experimental)
  Interventions: Drug: Fluzoparib with Temozolomide

INTERVENTIONS:
Drug: Fluzoparib with Temozolomide — Fluzoparib: 100mg, po.bid. Q4W, d1-28, for a total of 6 cycles
  Temozolomide (TMZ): 150-200 mg/m2, po. Q4W, d1-5, for a total of 6 cycles
  If unacceptable toxicity occurs and a dose reduction is required, it is recommended to first reduce the dose from 100 mg (2 tablets) to 50 mg (1 tablet) twice a day. If further dose reduction is required, it is recommended to reduce the dose from 50 mg (1 tablet) twice a day to 50 mg (1 tablet) once a day. If it is still intolerable, the patient should withdraw from the clinical study.
  The TMZ dose is adjusted by the investigator according to standard chemotherapy requirements. Adjuvant TMZ treatment of less than 6 cycles is allowed depending on the subject's condition (e.g. confirmed disease progression, intolerable toxicity, etc.). Tumor assessment is performed during two cycles of TMZ (q8w±7 days) during the study or when clinically indicated

SUMMARY:
A Phase II clinical study is planned to evaluate the efficacy and safety of fluzoparib combined with temozolomide in newly diagnosed glioblastoma patients after completing standard concurrent chemoradiotherapy (CCRT), explore the effectiveness and safety of this regimen, and find a better treatment option for glioblastoma patients

ELIGIBILITY:
Inclusion Criteria:

* 1.Signed informed consent form (ICF);

  2. Age ≥18 years old, <70 years old;

  3. Based on postoperative MRI, the total resection range is ≥80% compared with preoperative MRI (resection for the purpose of biopsy is not eligible);

  4. Patients newly diagnosed with primary glioblastoma by imaging or pathology, completed concurrent chemoradiotherapy (CCRT), and planned to receive adjuvant TMZ treatment;

  5. Appropriate hematological treatment and end-organ function within 14 days before randomization, defined by the following laboratory results:
  * Absolute neutrophil count (ANC) ≥1.5×109/L;
  * Platelet count ≥100×109/L;
  * Hemoglobin ≥90 g/L;
  * Total bilirubin ≤1.5 ×ULN;
  * AST and ALT ≤3 × ULN;
  * Alkaline phosphatase ≤2.5 × ULN;
  * Serum albumin ≥25 g/L;
  * Serum creatinine ≤133 μmol/L;
  * PT and aPTT ≤ 1.5 × ULN; 6. Karnofsky score ≥ 60; 7. Expected survival > 12 weeks; 8. Women of childbearing age*: must use highly effective contraceptive methods (resulting in a contraceptive failure rate of <1% per year) from the date of informed consent until at least 3 months after the last dose of the study drug fluzoparib/TMZ (whichever occurs later).

Men: agree to use contraceptive measures, defined as follows: For female partners of childbearing potential or pregnant female partners, men must use highly effective contraceptive methods from the date of informed consent until at least 3 months after the last dose of the study drug fluzoparib/TMZ (whichever occurs later).

*Women are postmenopausal women who have not reached postmenopausal status (continuous amenorrhea for ≥ 12 months without a confirmed cause other than menopause) and have not undergone surgical sterilization (removal of the ovaries and/or uterus).

Exclusion Criteria:

* 1. During the concurrent chemoradiotherapy phase, the total radiotherapy dose is >60Gy; 2. Multifocal glioma (≥3 lesions); 3. Patients with primary infratentorial glioblastoma; 4. Patients with leptomeningeal disease; 5. Patients with stable or no dose reduction of corticosteroids within 14 days of randomization; 6. Pregnancy, lactation or breastfeeding (need to breastfeed or breastfeed during the study);

  * Women of childbearing age (including women who have undergone tubal ligation) must undergo a blood pregnancy test 7. Major cardiovascular disease, including New York Heart Association heart disease (grade 2 or higher), myocardial infarction within 3 months before randomization, unstable arrhythmia requiring treatment within the first 3 months, and/or newly diagnosed unstable angina; 8. Known clinically significant liver disease, including active viral, alcoholic or other hepatitis, cirrhosis, and hereditary liver disease; 9. Poorly controlled type 2 diabetes, defined as glycated hemoglobin ≥8% or fasting blood glucose ≥8.8 during the screening period mmol/L; 10. Major surgery (requiring general anesthesia) is expected during the study; 11. Any severe or uncontrollable systemic disease, including uncontrollable hypertension (defined as blood pressure still higher than 150/90 mmHg after effective antihypertensive treatment) and active bleeding disorders; 12. Any anticancer treatment after CCRT, whether experimental or approved, including chemotherapy, immunotherapy, gene therapy, cancer vaccine, cell therapy, cytokine/hormone therapy, and/or radiotherapy; 13. Persistent toxicity related to previous treatment (according to NCI CTCAE v5.0 toxicity level as > 1); according to the investigator's judgment, alopecia, sensory neuropathy ≤ 2, or other safety risk level ≤ 2 are eligible for inclusion; 14. Malignant tumors other than the study disease within 5 years before randomization, except for patients without risk of death or metastasis (adequately treated cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer or ductal carcinoma in situ); 15. During the screening period, patients have active viral infections that require systemic treatment:

    * HIV antibody positive;
    * Active hepatitis B: defined as HBsAg positive or HBcAb positive, and HBV DNA test result > 2000 IU/mL;
    * Active hepatitis C: defined as HCV antibody positive and PCR test HCV RNA positive. However, subjects with positive serum anti-HCV and negative HCV RNA can also be included;
    * Syphilis infection (positive Treponema pallidum specific antibody); 16. Patients who the investigator believes are not suitable for participation in the trial or will violate the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
OS | Patients were assessed up to 36 months from enrollment to first death (whichever occurred first)
  Defined as the time from the date of randomization to death from any cause.

SECONDARY OUTCOMES:
PFS | From enrollment to the first appearance of disease progression or date death from any cause,whichever came first,assessed up to 36 mounths
  PFS is defined as the time (in days) from the first use of study drug to the first observation of disease progression.
ORR | From enrollment to initial efficacy evaluation ,assessed up to 6 months
  Objective response rate

IPD SHARING:
Plan to Share IPD: No